CLINICAL TRIAL: NCT02292745
Title: Efficacy and Feasibility of Combining FOLFIRINOX and Stereotactic Radiotherapy for Patients With Irresectable Locally Advanced Pancreatic Cancer.
Acronym: LAPC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014- 00235039; 2014-002350-39 (EudraCT Number)
Record Dates: First submitted 2014-07-28; First posted 2014-11-17 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Neoplasms
Keywords: locally advanced pancreatic cancer; chemotherapy; stereotactic radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic radiotherapy (Experimental): Standard of care FOLFIRINOX treatment followed by stereotactic radiotherapy
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: stereotactic radiotherapy

SUMMARY:
The purpose of this study is to investigate whether combining FOLFIRINOX chemotherapy and stereotactic radiotherapy in patients with locally advanced pancreatic cancer leads to an increase in survival.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histologically confirmation of pancreatic cancer.
* WHO performance status of 0 or 1
* ASA classification I or II
* Tumor considered locally advanced after diagnostic work-up including CT-imaging and diagnostic laparoscopy.
* No evidence of metastatic disease
* Largest tumor diameter < 7 cm x 7 cm x 7 cm
* Normal renal function (Creatinine ≥ 30 ml/min).
* Normal liver tests (bilirubin < 1.5 times normal; ALAT/ASAT < 5 times normal)
* Normal bone marrow function (WBC > 3.0 x 10e9/L, platelets > 100 x 10e9/L and hemoglobin > 5.6 mmol/l)
* Age > 18 years and < 75 years
* Written informed consent

Exclusion Criteria:

* Prior radiotherapy, chemotherapy or resection (bypass surgery allowed).
* Lymph node metastases from primary tumor outside the field of radiation.
* Second primary malignancy except in situ carcinoma of the cervix, adequately treated non-melanoma skin cancer, or other malignancy treated at least 3 years previously without evidence of recurrence.
* Pregnancy, breast feeding.
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 3.5 years after start of therapy

SECONDARY OUTCOMES:
number of toxicity events related to chemotherapy | up to 3.5 years after start of therapy
radiological response rates after chemotherapy and radiotherapy | up to 3.5 years after start of therapy
number of resections at end of stereotactic radiotherapy | up to 3.5 years after start of therapy
time to locoregional disease progression | up to 3.5 years after start of therapy
time to development of distant metastases | up to 3.5 years after start of therapy
predictive value of a set of biological markers for treatment response | up to 3.5 years after start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Prof. C.H.J. van Eijck, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Derived] Suker M, Nuyttens JJ, Eskens FALM, Haberkorn BCM, Coene PLO, van der Harst E, Bonsing BA, Vahrmeijer AL, Mieog JSD, Jan Swijnenburg R, Roos D, Koerkamp BG, van Eijck CHJ. Efficacy and feasibility of stereotactic radiotherapy after folfirinox in patients with locally advanced pancreatic cancer (LAPC-1 trial). EClinicalMedicine. 2019 Nov 19;17:100200. doi: 10.1016/j.eclinm.2019.10.013. eCollection 2019 Dec. PMID 31891135